CLINICAL TRIAL: NCT03676049
Title: Cannabidiol (CBD) Cannabis Extract Oral Solution for Drug Resistant Pediatric Epilepsy (Expanded Access Use)
Brief Title: Cannabidiol for Drug Resistant Pediatric Epilepsy (Expanded Access Use)
Status: Available | Type: Expanded Access
Sponsor: John (Other)
Responsible Party: Sponsor-Investigator, John, M.D., Associate Professor, University of Mississippi Medical Center
Organization: University of Mississippi Medical Center (Other)
Other Study IDs: 2017-0259
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Drug Resistant Epilepsy
Keywords: Children, Epilepsy, Cannabidiol
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Cannabidiol — CBD will be administered as an adjunct to all current antiepileptic drugs. A dosing titration period will start with 100 mg/day, with 50mg BID dosing, and will be titrated monthly as tolerated based on clinical response, up to 300mg/day. This is based on a targeted dosing of 2.5 ---5---7.5 mg/kg/d.
  Other Names: CBD

SUMMARY:
This is a treatment study under an approved Expanded Use IND protocol for using Cannabidiol (CBD) Extract. CBD will be used for the treatment of 5-10 children with drug resistant epilepsy. The CBD used in this study is prepared at the University of Mississippi under approval of the National Institute on Drug Abuse (NIDA) for its preparation and FDA approval under an expanded access mechanism on a compassionate use basis. The target patient population is who would otherwise have no appropriate remaining treatment modality left. These are patients for whom the risks of a relatively untested product are outweighed by the potential benefit. Using seizure-diaries to register seizure frequency, drug log and questionnaire to measure parent/patient quality of life and side effects will be assessed in each visit. Visits are: baseline, 4, 8, and 12 weeks visit. A 24 weeks visit (6 months) will be performed if the patient is stable on therapy during the 3 initial months and want to continue on the study for 3 more months. CBD will be administered as an adjunct to all current anti-epileptic therapies.

DETAILED DESCRIPTION:
Expanded Access Use: Restrictions to those with most significant epilepsy severity and especially neurocognitive delays (to minimize side effect profiles) remain in place. Study design, hover, is targeted at an Expanded Access use of product for children who would otherwise have no appropriate remaining treatment modality left.

Timeline: 3 months with the option to continue for up to 3 months of follow up therapy.

Procedures:

Participants: Five to ten (5-10) refractory epilepsy patients, aged 5-19 years old, all sexes, who must have failed at least 3 appropriate drugs, +/- vagal nerve stimulator, +/- dietary therapy, +/- resective surgery will be provided CBD as part of the Principal Investigator's Physician Expanded Access IND.

Written parental permission obtained from the patient's parent or legal representative must be obtained prior to beginning treatment.

Drug administration: CBD will be administered as an adjunct to all current antiepileptic drugs. A dosing titration period will start with 100 mg/day, with 50mg BID dosing, and will be titrated monthly as tolerated based on clinical response, up to 300mg/day. This is based on a targeted dosing of 2.5---5---7.5 mg/kg/d. Any patients under 40kg will have adjusted dosing based on weight as follows:

For 40 kg and up:

1 ml BID, escalating to 2 ml BID, and then 3 ml BID

For 30 - 39 kg:

0.75 ml BID, escalating to 1.5 and 2.25 ml BID

For 20 - 29 kg 0.5 ml BID, escalating to 1 and 1.5 ml BID

Clinical evaluations: All subjects will be clinically evaluated at baseline, once a month for the three months of titration period and during the three months of follow up period. During the first week of the study drug initiation, patients will be called at day 3 and then at day 7 to review any changes in condition. Subsequently, patients will receive a phone call weekly and will be evaluated in their physician study visits during the titration period to review any changes in condition and determine whether an increase in dosing is required. The investigator will be available by telephone throughout the 3 months of the titration period of the study, in between the visits and throughout the 3 months in the follow up period. Patients will receive the CBD during their monthly study visits during the titration and follow up period. The first dose of CBD will be administered by the physician in the Pediatric Clinical Research Clinic.

Pregnant patients will be excluded from the study. Female patients of childbearing potential will be screened for pregnancy prior to enrollment, and during the study if a potential for pregnancy arise. A -blood pregnancy test will be used. Therefore, parent/guardian of female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if the child become pregnant during the study.

During the study, the patients will be constantly monitored as the investigators describe below:

Onset:

* Pediatric Neurology Physician evaluation.
* Initial lab work to include complete blood counts, comprehensive metabolic panel and baseline co-existent antiepileptic drug levels. Blood pregnancy testing will be performed on those patients with childbearing potential.
* Initial body weight and routine vital signs
* Initial baseline Electroencephalogram (EEG). Video EEG prior to enrollment if epileptic syndrome or severity is unclear. Decision and enrollment classification to be made by Dr. Ingram prior to enrollment.
* Patient quality of life, side effect profile, and seizure count will be completed as typical clinical interview prior to enrollment.

  4 weeks/1 month:
* Pediatric Neurology Physician evaluation.
* Lab work to include complete blood counts, comprehensive metabolic panel and concomitant epilepsy medication levels. Blood testing for CBD/THC will also be performed. Additional lab draws can be performed with any symptoms to suggest anticonvulsant toxicity or concerning clinical signs/symptoms.
* Patient quality of life, side effect profile, and seizure count will be completed as typical clinical interview at the end of 1-month study window.

  8 weeks/2 months:
* Pediatric Neurology Physician evaluation.
* Lab work as indicated for 4 weeks/1 month.
* Body weight and routine vital signs
* Patient quality of life, side effect profile, and seizure count will be completed as typical clinical interview at the end of 2-months study window.

  12 weeks/3 months:
* Pediatric Neurology Physician evaluation.
* EEG at the completion of the 3-month study window.
* Lab work as indicated for 4 weeks/1 month.
* Body weight and routine vital signs
* Patient quality of life, side effect profile, and seizure count will be completed as typical clinical interview at the end of 3-months study window.

Follow up:

Patients who are stable on therapy and happy with the results may remain on study for up to 3 more months after titration period. These patients will have 6 months total on medication and one visit/month during the follow up time for clinical evaluation:

* Complete blood count
* Comprehensive metabolic profile (including liver function tests)
* Measurement of levels of concomitant anti-epileptic drugs
* Patient quality of life, side effect profile, and seizure count will be completed as typical clinical interview.
* EEG (at 6 months visit)

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria will be considered eligible for this study:

* Age 5-19 years old
* Documentation of a diagnosis of drug resistance epilepsy as evidenced by failure to control seizures despite appropriate trial of three or more anti-epileptic drugs at therapeutic doses. Some of these drugs include Brivaracetam, Carbamazepine, Clobazam, Clonazepam, Diazepam, Divalproex Sodium, Eslicarbazepine Acetate, Ethosuximide, Felbamate, Gabapentin, Lacosamide, Lamotrigine, Levetiracetam, Lorazepam, Oxcarbazepine, Perampanel, Phenobarbital, Phenytoin, Pregabalin, Rufinamide, Valproic Acid, Vigabatrin, Zonisamide. Documentation must include the diagnosis of epilepsy type or epilepsy syndrome (if possible), as well as the underlying case, when known.
* Between 1-3 baseline anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment. Vagus nerve stimulator, and dietary therapies do not count toward this parameter, but are not bases for exclusion.
* Vagus nerve stimulator must be on stable settings for a minimum of 3 months.
* A history of significant epilepsy severity and neurocognitive delays, specifically a baseline history of being nonverbal and non-ambulatory without assistance

Exclusion Criteria:

The patient may not enter the study if ANY of the following apply:

* Patients with resectable epilepsy or syndromes where dietary or other therapy is first line will not be enrolled prior to attempting those therapies with failure OR parental refusal of said therapies.
* Treatment with any artisanal preparation containing or possible containing CBD during the month before initiation of the study drug.
* Allergy to CBD or any cannabinoid.
* Unable to comply with study visits/requirements.
* CBD is contraindicated in pregnancy and during breast-feeding. Female subjects who are pregnant or breastfeeding will be excluded from treatment with CBD. Patients of childbearing potential will be screened for pregnancy prior to enrollment and during the study if a potential for pregnancy arise. A blood pregnancy test will be used. Additionally, for patients of childbearing potential, enrollment criteria will require the use of highly effective contraception (e.g. double barrier, abstinence, or IUD) for the duration of treatment with CBD. Therefore, parent/guardian of female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if the child become pregnant during the study.
* Significant impaired hepatic function at screening as characterized by one of the following:

  i. Alanine aminotransferase [ALT] >5 × upper limit of normal (ULN) and total bilirubin (TBL) >2 × ULN ii. ALT or Aspartate aminotransferase (AST) >3 × ULN and either TBL >2 × ULN or international normalized ratio (INR) >1.5
* History or presence of alcohol or substance abuse
* Use of other cannabis or CBD products

Ages: 5 Years to 19 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States